CLINICAL TRIAL: NCT03570151
Title: Medical Care at a Mass-gathering Music Festival: A Retrospective Study Over Seven Years (2011 - 2017) of the Frequency Festival
Brief Title: Medical Care at a Mass-gathering Music Festival
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Mathias Maleczek, Principal investigator, Medical University of Vienna
Other Study IDs: FRQ
Record Dates: First submitted 2018-06-15; First posted 2018-06-26 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: All Health Problems Occurring During a Music Festival

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention will be done

SUMMARY:
Key Objective is to describe Patient Presentation Rate and Transport to Hospital rate at an Austrian Music Festival. If significant changes in specific incidence rates are found, a causal explanation will be looked for.

ELIGIBILITY:
Inclusion Criteria:

* All persons seeking help from the local ambulance service at the music festival

Exclusion Criteria:

* Incomplete Data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Visitors and staff at an Austrian music festival
Sampling Method: Probability Sample
Enrollment: 18684 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Patient Presentation Rate | 2011-2017
  Patients per 1000 visitors
Transfer to Hospital Rate | 2011-2017
  Hospitalisations per 1000 visitors

SECONDARY OUTCOMES:
Changes in the Incidence of single Illnesses | 2011-2017

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No